CLINICAL TRIAL: NCT04922112
Title: Sleep Apnea in Head and Neck Cancer Patients at the University of Colorado
Acronym: OSA-HN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to find participants, no enrollment
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-1778.cc; P30CA046934 (NIH)
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Obstructive Sleep Apnea; Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Sleep Apnea, Obstructive; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Research group (Experimental): Sleep apnea testing will be performed with this group, in the form of quality of life and sleep questionnaires, home sleep study results, as well as information collected from their electronic medical record. The investigator will also obtain blood laboratory specimens to measure serum TNF-alpha and IL-6.
  Interventions: Diagnostic Test: Obstructive sleep apnea testing

INTERVENTIONS:
Diagnostic Test: Obstructive sleep apnea testing — * Functional Outcomes of Sleep Questionnaire (FOSQ-10)
  * European Organization for Research and Treatment of Cancer Head and Neck Survey (EORTC HN 35)
  * Epworth Sleepiness Scale (ESS)
  * Adult Comorbidity Evaluation (ACE 27)
  * University of Washington Quality of Life Questionnaire (UW-QOL)
  * Chronic Pain Assessment Questionnaire

SUMMARY:
Obstructive sleep apnea (OSA) is increasingly recognized in patients with squamous cell carcinoma of the head and neck (SCCHN). The prevalence prior and after cancer therapy is not well understood. OSA is identified as a contributing factor for daytime somnolence and quality of life (QOL), yet treatment of OSA in the SCCHN population has not been studied. The investigators hope to identify the disease course of sleep apnea, risk factors for development, and impact on QOL with treatment of OSA in a population of patients with SCCHN.

DETAILED DESCRIPTION:
The investigators will conduct a prospective cohort study of enrolled patients seen in initial consultation by our H&N cancer surgeons and/or Radiation Oncologists either at AMC or HRH. Data collected from patients in the form of quality of life and sleep questionnaires and home sleep study (Alice Night One System by Phillips Respironics), as well as data from the electronic medical record will be coded into RedCap.

Blood collection for inflammatory biomarkers will occur during routine laboratory workup to avoid unnecessary phlebotomy whenever possible. Blood laboratory specimens of the inflammatory markers will be centrifuged to plasma and stored at -80C in freezers located on the Anschutz campus in Research Complex 2 on the 7th floor. Patients who require tracheostomy will be included in this study but will not have any sleep study time-point as indicated. Patients who are identified to have OSA will undergo counseling and treatment as per standard of care. CPAP compliance data will be collected every three months after initiation of OSA treatment.

Patient details including demographics, treatment information such as surgery, radiation, and chemotherapy, sleep and quality of life questionnaire data, pro-inflammatory cytokines, and sleep study results will collected. The RedCap database will be maintained by the PI, or their delegate of the present study, and all persons utilizing the RedCap database for purposes of entering data will be included on the Delegation of Authority.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between the ages of 21 (inclusive) and 90 (inclusive). Anyone that is over 89 years old will be labeled as 89 in the data analysis.
2. Patients with an established relationship with the adult Otolaryngology and/or Radiation Oncology clinic at AMC or HRH.
3. Patients that present with a new diagnosis of oropharyngeal SCC who undergo radiation treatment, with or without chemotherapy.
4. Patients who may require trachesotomy will be included.
5. Stated willingness to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

1. Under the age of 21 or over the age of 90.
2. Unwilling to sign the informed consent.
3. Unable or unwilling to participate in sleep studies.
4. Patients who have had a prior diagnosis of SCCa of the head and neck including nasopharynx, oral cavity, oropharynx, larynx and hypopharynx will be excluded. Patients with prior non-cutnaeous non-SCC tumors of the head and neck will also be excluded. Patients with prior skin cancer diagnoses will not be excluded.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
FOSQ-10 (Functional Outcomes of Sleep Questionnaire) | 72 weeks
  Measurement of daytime somnolence impact on activities of daily living. Score 0-4 for each item, with a score range of 5-20, higher scores with better outcome
EORTC-HN35 (European Organization for Research and Treatment of Cancer) | 72 weeks
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-QLQ-H&N35. Qquality of life assessment in head and neck cancer patients. A raw score is calculated as a mean of the component items, then a linear transformation is performed with score of 0 to 100; the summary score is an average of the raw scores of each group of questions. A higher scores indicate greater impairment.
ESS (Epworth Sleepiness Scale) | 72 weeks
  A measure of daytime sleepiness. Score 0-4 for each item, score range 0-24, higher scores with worse outcome.
ACE-27 (Adult Comorbidity Evaluation 27) | 72 weeks
  Comorbidity instrument/severity. Score 0-3 with higher scores with worse outcome.
UW-QOL (University of Washington Quality of Life Questionnaire) | 72 weeks
  Provides basic quality of life data on the physical, functional, emotional quality of life of the head and neck cancer patient. Score 0-100 with the higher score the better outcome.
Chronic Pain Assessment | 72 weeks
  Assess chronic pain that changes over time, persistent baseline and breakthrough pain. This isn't scored in the same way, but the severity of pain scale 0-10 and use of medications will be compared. A higher score is worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No